CLINICAL TRIAL: NCT07268248
Title: 1-hour Premedication for Allergy Goal in Emergency Computed Tomography, A Multicenter Randomized Controlled Non-inferiority Trial: PAGE-1 Study
Brief Title: 1-hour Premedication for Allergy Goal in Emergency: PAGE-1 Study
Acronym: PAGE1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Peng, MD PhD MSCR (Other)
Responsible Party: Sponsor-Investigator, Paul Peng, MD PhD MSCR, Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2025002416
Record Dates: First submitted 2025-11-21; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Allergic Reaction to Contrast Media; Hypersensitivity Reaction; Computed Tomography; Premedication
Keywords: Iodinated Contrast Reaction; Contrast-enhanced CT; Glucocorticoid prophylaxis
MeSH Terms: conditions — Hypersensitivity | interventions — Glucocorticoids; Histamine Antagonists; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-hour Premedication Protocol (Experimental): IV glucocorticoid and antihistamine 1 hour before contrast
  Interventions: Other: IV glucocorticoid and antihistamine
- 4-hour Premedication Protocol (Active Comparator): IV glucocorticoid 4 hours before contrast and IV antihistamine 1 hour before contrast
  Interventions: Other: IV glucocorticoid and antihistamine (standard of care)

INTERVENTIONS:
Other: IV glucocorticoid and antihistamine — Methylprednisolone sodium succinate (e.g., Solu-Medrol®) 40 mg IV immediately plus diphenhydramine 25 mg IV 1 hour before contrast medium administration for CT imaging
  Arms: 1-hour Premedication Protocol
Other: IV glucocorticoid and antihistamine (standard of care) — Methylprednisolone sodium succinate (e.g., Solu-Medrol®) 40 mg IV immediately 4 hours before contrast medium administration, plus diphenhydramine 25 mg IV 1 hour before contrast for CT imaging
  Arms: 4-hour Premedication Protocol

SUMMARY:
1-hour Premedication for Allergy Goal in Emergency: PAGE-1 is a prospective, parallel, two-arm, non-inferiority, multicenter randomized controlled trial evaluating the safety of a 1-hour (intervention) versus a 4-hour (standard regimen) intravenous (IV) premedication protocol in adult patients in the Emergency Department (ED) with a documented iodinated contrast allergy and requiring computed tomography (CT) imaging for a high-risk indication.

DETAILED DESCRIPTION:
Allergic or hypersensitivity reactions to iodinated contrast media are rare, estimated to occur in 0.3% to 1.4% of cases, but have decreased significantly after the switch from high-osmolar to low-osmolar contrast. Most reactions are mild, and breakthrough reactions occur regardless of the timing of premedication. IV premedication is recommended, but there is no level I evidence for its basis in the ED.

This study addresses the sparse evidence that underpins the ubiquitous multi-hour premedication protocols in EDs nationwide. It specifically challenges the existing paradigm of 4-5 hours of IV premedication, which has remarkably never been prospectively validated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 21 years old)
2. Documented iodinated contrast allergy in the electronic health record
3. CT with iodinated contrast ordered for a high-risk indication, † defined as post-arrest, concern for aortic dissection, ischemia, occlusion, obstruction, or other life-threatening conditions requiring timely diagnosis
4. Willing and able to give consent

Exclusion Criteria:

1. Previous enrollment in this study
2. Pregnancy
3. Seafood or iodine allergy, alone
4. Gadolinium allergy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of Acute Contrast Reaction | 30 minutes
  Measurement of any contrast reaction after contrast administration
Proportion of patients eligible for intervention | Before randomization
  Ratio of those eligible to screened

SECONDARY OUTCOMES:
Proportion randomized to intervention and control | Within 30 minutes after completion of CT imaging
  Ratio of patients randomized to intervention and control arms, and who complete the protocol as specified
Adverse events after intervention | Within 30 minutes after assessment of primary outcome
  Proportion of patients who required intramuscular epinephrine, noninvasive ventilation, or intubation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Peng, Principal Investigator — Rutgers Robert Wood Johnson Medical School

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical plan
Supporting Information: Study Protocol, SAP
Time Frame: Available after start date and 1 year after end of study
Access Criteria: Study coordinators and key personnel
URL: http://redcap.rutgers.edu

REFERENCES:
- [Background] Davenport MS, Cohan RH. The Evidence for and Against Corticosteroid Prophylaxis in At-Risk Patients. Radiol Clin North Am. 2017 Mar;55(2):413-421. doi: 10.1016/j.rcl.2016.10.012. PMID 28126223
- [Background] Greenberger PA, Halwig JM, Patterson R, Wallemark CB. Emergency administration of radiocontrast media in high-risk patients. J Allergy Clin Immunol. 1986 Apr;77(4):630-4. doi: 10.1016/0091-6749(86)90357-x. PMID 3958391
- [Background] Lasser EC, Berry CC, Talner LB, Santini LC, Lang EK, Gerber FH, Stolberg HO. Pretreatment with corticosteroids to alleviate reactions to intravenous contrast material. N Engl J Med. 1987 Oct 1;317(14):845-9. doi: 10.1056/NEJM198710013171401. PMID 3627208
- [Background] Katayama H, Yamaguchi K, Kozuka T, Takashima T, Seez P, Matsuura K. Adverse reactions to ionic and nonionic contrast media. A report from the Japanese Committee on the Safety of Contrast Media. Radiology. 1990 Jun;175(3):621-8. doi: 10.1148/radiology.175.3.2343107.
- [Background] Amiri E. Optimizing Premedication Strategies for Iodinated Contrast Media in CT scans: A Literature Review. J Med Imaging Radiat Sci. 2025 Jan;56(1):101782. doi: 10.1016/j.jmir.2024.101782. Epub 2024 Nov 20. PMID 39571411
- [Background] Freed KS, Leder RA, Alexander C, DeLong DM, Kliewer MA. Breakthrough adverse reactions to low-osmolar contrast media after steroid premedication. AJR Am J Roentgenol. 2001 Jun;176(6):1389-92. doi: 10.2214/ajr.176.6.1761389. PMID 11373198
- [Background] Mervak BM, Davenport MS, Ellis JH, Cohan RH. Rates of Breakthrough Reactions in Inpatients at High Risk Receiving Premedication Before Contrast-Enhanced CT. AJR Am J Roentgenol. 2015 Jul;205(1):77-84. doi: 10.2214/AJR.14.13810. PMID 26102383
- [Background] Mervak BM, Cohan RH, Ellis JH, Khalatbari S, Davenport MS. Intravenous Corticosteroid Premedication Administered 5 Hours before CT Compared with a Traditional 13-Hour Oral Regimen. Radiology. 2017 Nov;285(2):425-433. doi: 10.1148/radiol.2017170107. Epub 2017 Jul 26. PMID 28745940
- [Background] Wang CL, Cohan RH, Ellis JH, Caoili EM, Wang G, Francis IR. Frequency, outcome, and appropriateness of treatment of nonionic iodinated contrast media reactions. AJR Am J Roentgenol. 2008 Aug;191(2):409-15. doi: 10.2214/AJR.07.3421. PMID 18647910
- [Background] Goldfarb JW. National trends in contrast media enhanced and unenhanced computed tomography use. Clin Imaging. 2023 Jan;93:103-105. doi: 10.1016/j.clinimag.2022.11.009. Epub 2022 Nov 17. No abstract available. PMID 36427426
- [Background] Berlyand Y, Fraga JA, Succi MD, Yun BJ, Lee AH, Baugh JJ, Whitehead D, Raja AS, Prabhakar AM. Impact of iodinated contrast allergies on emergency department operations. Am J Emerg Med. 2022 Nov;61:127-130. doi: 10.1016/j.ajem.2022.08.052. Epub 2022 Sep 5. PMID 36096014
- [Background] Wang C, Ramsey A, Lang D, Maria Copaescu A, Krishnan P, Kuruvilla M, Mervak B, Newhouse J, Sumkin A, Saff R. Management and Prevention of Hypersensitivity Reactions to Radiocontrast Media: A Consensus Statement from the American College of Radiology and the American Academy of Allergy, Asthma & Immunology. Radiology. 2025 May;315(2):e240100. doi: 10.1148/radiol.240100. PMID 40326871